CLINICAL TRIAL: NCT07228936
Title: Evaluation of the Association Between Pectoralis Minor Tightness and the Initiation Site of Rotator Cuff Tears: A PRospective Single Center Observational Study
Brief Title: Association of Pectoralis Minor Tightness With the Initiation Site of Rotator Cuff Tears
Acronym: PMinor-Rotator
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagatay Delice, STUDY_CHAİR GAZİ UNİVERSİTY, Gazi University
Other Study IDs: E-77082166-302.08.01-1273486
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Impingement Syndrome; Rotator Cuff Injuries; Pectoralis Minor Tightness; Pectoralis Minor Muscle Tension
Keywords: rotator cuff; Rotator Cuff Injuries; Posture; Scapula; Pectoralis Muscles; Arthroscopy; Shoulder Joint; Pectoralis Minor
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at whether tightness of a small chest muscle called the pectoralis minor is linked to where rotator cuff tears begin in the shoulder. Rotator cuff tears can start on the bursal side (top surface) or the articular side (joint surface). We want to learn if people with a tighter pectoralis minor are more likely to have tears that begin on the bursal side.

Adults aged 18-60 who already plan to have shoulder arthroscopy as part of their usual medical care at Gazi University Hospital may be invited. Taking part does not change their treatment. Before surgery, a trained clinician will measure shoulder posture and pectoralis minor length using simple external tools (a caliper and ruler-like square). We will also review routine shoulder X-rays and MRI scans if available. During surgery, the surgeon will look inside the joint (standard arthroscopy) and record where the tear appears to start. No extra procedures are added for research.

We expect to include about 81 participants. The main question is whether people with a shorter (tighter) pectoralis minor more often have bursal-side tear initiation. Results may help doctors understand shoulder mechanics and improve prevention or rehabilitation strategies in the future. Participation is voluntary, and data will be de-identified and kept confidential. There is no direct benefit to participants, and risks are limited to the brief, noninvasive measurements performed before surgery.

DETAILED DESCRIPTION:
Detailed Description

Rationale and Objectives Pectoralis minor (PM) tightness alters scapular position (anterior tilt, internal rotation) and may increase subacromial compression. This study prospectively evaluates whether PM tightness is associated with the initiation site of rotator cuff tears (RCTs)-specifically, whether tears more often begin on the bursal side in shoulders with a shorter (tighter) PM.

Design and Setting Single-center, prospective, observational study at a tertiary academic hospital (orthopaedic shoulder service). Care is not altered by participation. All surgical and imaging procedures are standard of care; research procedures are limited to noninvasive postural/PM length measurements and structured data collection.

Participants Adults scheduled for routine shoulder arthroscopy for suspected/confirmed RCT may be invited. Key exclusions (summarized): prior ipsilateral shoulder surgery; acute fracture/dislocation; major-trauma RCT; cervical radiculopathy/thoracic outlet syndrome; systemic inflammatory arthropathy; barriers to consent. (Full inclusion/exclusion are listed in the Eligibility section.)

Study Procedures

Preoperative assessments (same-day or pre-op clinic):

Pectoralis minor length (mm): Linear distance from coracoid tip to rib attachment measured with a digital caliper; three trials recorded; mean used for analysis.

Scapular posture metrics:

Medial scapular border-thoracic distance (mm) using calipers/ruler. Forward shoulder posture using a 300 mm square/ruler referenced to the table/chest wall.

Imaging abstraction: Standard shoulder radiographs and MRI summarized (tear size/pattern, fatty infiltration grades if reported).

Intraoperative assessment (standard arthroscopy):

Surgeons document tear initiation site (bursal vs articular/delamination) and tear characteristics (pattern/size) using a standardized form based on video visualization. No additional portals or procedures are performed for research.

Data Elements and Sources

Source documents: medical records, PACS (X-ray/MRI), operative reports, arthroscopy video, and study case report forms (CRFs).

Key variables: PM length (continuous, mm); posture measures; tear initiation site (primary outcome); tear size/pattern; demographic/clinical covariates (age, sex, side, symptom duration, occupation/sport, BMI if available).

Registry Operations and Quality Plan

Quality Assurance & Monitoring

Training/standardization: Investigators receive a 1-page landmarking guide and a brief hands-on calibration session for PM and scapular measurements.

Inter-/intra-rater reliability: A random 15-patient subset will be re-measured by a second rater within the same visit; intraclass correlation coefficients (ICC, two-way random, absolute agreement) will be reported.

Instrument calibration: Digital calipers checked weekly with a gauge block; records kept in a calibration log.

On-site checks: Monthly coordinator audits of 10% of charts for consent presence, eligibility, and CRF completeness.

Automated Data Checks

Electronic CRFs include range checks (e.g., PM length 80-200 mm; posture distances 0-100 mm) and logic checks (e.g., surgery date ≥ consent date; side consistency across forms).

Cross-field consistency rules (examples): if "tear initiation = bursal," then arthroscopy notes must include bursal-surface description; MRI "no tear" triggers manual review of intraop outcome.

Source Data Verification (SDV)

100% SDV of primary outcome (tear initiation site) against operative video/report.

20% SDV of key predictors (PM length, posture metrics) against paper measurement sheets.

Discrepancies >2 mm or any categorical mismatch prompt corrective action and retraining as needed.

Data Dictionary

A structured dictionary defines each variable (name, label, unit, allowed values, derivation, normal/expected range, source document, and coding system where relevant-e.g., MedDRA for adverse events).

Versioned and stored with the analysis code; any change triggers a minor version update and change log entry.

Standard Operating Procedures (SOPs) SOPs cover: screening and consent; measurements; data entry; query resolution; SDV/monitoring; adverse-event reporting (see below); database lock and change management; archiving and access control.

Sample Size and Power

Based on a logistic-regression framework with the primary outcome "bursal-side initiation (yes/no)," assumptions were: α=0.05 (two-sided), power=0.80, baseline bursal-initiation proportion ~0.50, prevalence of PM tightness ~0.50, and an odds ratio of ~4.0 for PM-tight vs non-tight. Variance-adjusted calculations support ≈82 shoulders total, satisfying ≥10 events per predictor for the planned model.

Plan for Missing Data

Prevention: required-field checks at data entry; real-time prompts for missing or out-of-range values.

Handling: if ≤5% missing for a covariate, complete-case analysis will be used; if >5-20%, single-variable multiple imputation (m = 20) under missing-at-random assumptions will be applied for predictors (not for outcomes). Sensitivity analyses will compare imputed vs complete-case results.

Outcome data: primary outcome (tear initiation site) is expected to be complete; any missing outcome leads to exclusion from the primary analysis and description of reasons.

Statistical Analysis Plan (SAP)

Descriptive analysis: Means/SD or medians/IQR for continuous variables; counts/percentages for categorical variables. Group summaries by PM-tight vs non-tight may be shown for context.

Primary analysis: Binary logistic regression with tear initiation site (bursal=1, articular/delamination=0) as the dependent variable; key predictor is PM length (continuous, per-10 mm decrease) and/or PM-tightness (binary, threshold prespecified from literature or study distribution).

Covariate adjustment: Age, sex, side, tear size/pattern, acromial morphology, and other prespecified clinical factors if available.

Model diagnostics: Linearity (Box-Tidwell for continuous predictors), multicollinearity (VIF<5), calibration (Hosmer-Lemeshow), discrimination (AUC with 95% CI).

Sensitivity analyses: (1) Treat PM length as continuous vs categorical; (2) exclude massive tears; (3) rater-blinded subset; (4) alternative PM-tightness cut-points (±5 mm).

Significance level: two-sided α=0.05 with 95% CIs; no multiplicity adjustment for the single primary endpoint.

Safety/Adverse Events

No investigational procedures are performed. The physical measurements are brief, external, and low-risk (possible transient discomfort). Any adverse events observed in proximity to research procedures will be recorded and reported per institutional policy. Surgical complications are part of routine care and will be documented but not attributed to research unless clearly related to the measurement process.

Data Management, Confidentiality, and Access

Data are recorded on coded CRFs and stored in a secure, access-controlled database. A link file that maps codes to identities is stored separately on encrypted drives. Access is role-based (PI, coordinator, analyst). Backups occur daily. Data retention follows institutional policy and national data-protection law.

Dissemination/IPD Sharing: Results will be submitted for publication and conference presentation. De-identified dataset and analysis code may be shared upon reasonable request after publication, subject to applicable privacy regulations and approvals.

Timeline: Anticipated start and completion dates match the Ethics approval window; enrollment begins only after registration posting and Ethics approval confirmation.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 60 years old.
* Shoulder pain.
* Suspected or confirmed rotator cuff tear by exam and/or imaging.
* Scheduled for shoulder arthroscopy as part of usual care.
* Willing to take part and give informed consent.

Exclusion Criteria:

* Previous surgery on the same shoulder.
* Recent traumatic shoulder injury such as fracture or dislocation.
* Rotator cuff tear due to major trauma.
* Neck/nerve conditions affecting the shoulder, such as cervical radiculopathy or thoracic outlet syndrome.
* Systemic inflammatory joint disease, such as rheumatoid arthritis or ankylosing spondylitis.
* Cognitive or communication problems that would prevent accurate measurements or consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients receiving care at a tertiary orthopaedic shoulder service (Gazi University Hospital, Ankara, Türkiye). Participants will be drawn from the hospital's outpatient clinics and scheduled surgical lists for shoulder arthroscopy, reflecting the routine referral/catchment population of the region. Consecutive eligible patients will be approached during preoperative visits.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Tear initiation site (Bursal, Articular, Delamination) | Intraoperative, Day 0 (index arthroscopy)
  Arthroscopic classification of the surface on which the rotator cuff tear appears to begin (bursal; articular/delamination), recorded with a standardized intraoperative checklist. Primary analysis: association between pectoralis minor (PM) length and bursal-side initiation (logistic regression; effect per 10-mm decrease in PM length and/or PM-tight vs non-tight).

SECONDARY OUTCOMES:
Pectoralis minor length | Preoperative assessment, Day 0
  Linear distance (mm) from coracoid tip to rib attachment site measured with a digital caliper; three trials (mean used for analysis). Reliability assessed statistically.
Forward shoulder posture | Preoperative assessment, Day 0
  Anterior displacement of the acromion relative to the thorax measured with a square ruler (standardized upright position). Three trials; mean used.
Medial Scapular Border Thoracic Distance | Preoperative assessment, Day 0
  Periscapular prominence measured with calipers at the medial scapular border in standardized upright posture; three trials, mean used.
Thoracic Kyphosis (Cobb angle) | Preoperative imaging review, Day 0
  Lateral thoracic radiograph measured using the Cobb method: superior endplate line of T5 and inferior endplate line of T12 (use closest visible end vertebrae if either is obscured). Lines perpendicular to each endplate are drawn; the included angle is recorded as the thoracic kyphosis Cobb angle. One trained assessor performs the measurement; a second assessor repeats it in a 15-case subset for reliability.
Scapular index (Coracoid-Sternum/Acromian lateral tip - thoracic spine) | Preoperative assessment, Day 0
  Ration of two linear distances measured with a digital caliper in standardized upright posture arms relaxed at sides.
  1. Coracoid-Sternum (mm) : shortest straight-line distance from the coracoid tip to the midline of the sternum at the manubrium level.
  2. Acromian lateral tip - Thoracic spine: straight-line distance from the most lateral point of the acromion to the tip of the thoracic spine.
  Scapular Index = (Coracoid-Sternum) / (Acromion- Thoracic spine). Three trials per shoulder; the mean ratio is used for analysis. A 15-case subset will be re-measured by a second rater to assess inter-rater reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Hospital, Ankara, Cankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Oyama S, Myers JB, Wassinger CA, Daniel Ricci R, Lephart SM. Asymmetric resting scapular posture in healthy overhead athletes. J Athl Train. 2008 Oct-Dec;43(6):565-70. doi: 10.4085/1062-6050-43.6.565. PMID 19030133
- [Background] Borstad JD, Ludewig PM. The effect of long versus short pectoralis minor resting length on scapular kinematics in healthy individuals. J Orthop Sports Phys Ther. 2005 Apr;35(4):227-38. doi: 10.2519/jospt.2005.35.4.227. PMID 15901124
- [Background] Ludewig PM, Reynolds JF. The association of scapular kinematics and glenohumeral joint pathologies. J Orthop Sports Phys Ther. 2009 Feb;39(2):90-104. doi: 10.2519/jospt.2009.2808. PMID 19194022
- [Background] Cools AM, Struyf F, De Mey K, Maenhout A, Castelein B, Cagnie B. Rehabilitation of scapular dyskinesis: from the office worker to the elite overhead athlete. Br J Sports Med. 2014 Apr;48(8):692-7. doi: 10.1136/bjsports-2013-092148. Epub 2013 May 18. PMID 23687006
- [Background] Yamaguchi K, Ditsios K, Middleton WD, Hildebolt CF, Galatz LM, Teefey SA. The demographic and morphological features of rotator cuff disease. A comparison of asymptomatic and symptomatic shoulders. J Bone Joint Surg Am. 2006 Aug;88(8):1699-704. doi: 10.2106/JBJS.E.00835. PMID 16882890
- [Background] Kibler WB, McMullen J. Scapular dyskinesis and its relation to shoulder pain. J Am Acad Orthop Surg. 2003 Mar-Apr;11(2):142-51. doi: 10.5435/00124635-200303000-00008. PMID 12670140
- [Background] Peterson DE, Blankenship KR, Robb JB, Walker MJ, Bryan JM, Stetts DM, Mincey LM, Simmons GE. Investigation of the validity and reliability of four objective techniques for measuring forward shoulder posture. J Orthop Sports Phys Ther. 1997 Jan;25(1):34-42. doi: 10.2519/jospt.1997.25.1.34. PMID 8979174
- [Background] Du WY, Huang TS, Hsu KC, Lin JJ. Measurement of scapular medial border and inferior angle prominence using a novel scapulometer: A reliability and validity study. Musculoskelet Sci Pract. 2017 Dec;32:120-126. doi: 10.1016/j.msksp.2017.08.004. Epub 2017 Aug 15. PMID 28827031
- [Background] Borstad JD. Measurement of pectoralis minor muscle length: validation and clinical application. J Orthop Sports Phys Ther. 2008 Apr;38(4):169-74. doi: 10.2519/jospt.2008.2723. Epub 2007 Nov 21. PMID 18434665